CLINICAL TRIAL: NCT05493514
Title: Clinical and Instrumental Treatment's Predictors in Subjects With Neurological Diseases Using G-EO Robotic System: an Observational Longitudinal Study
Brief Title: Clinical and Instrumental Treatment's Predictors in Subjects With Neurological Diseases Using G-EO Robotic System
Status: Recruiting | Type: Observational
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Responsible Party: Sponsor
Other Study IDs: 03_06/04/2022
Record Dates: First submitted 2022-07-21; First posted 2022-08-09 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-06

CONDITIONS: Multiple Sclerosis; Stroke; Parkinson Disease; Acquired Brain Injury
Keywords: Multiple Sclerosis; Stroke; Parkinson Disease; Acquired Brain Injury; Robotic; End-effector
MeSH Terms: conditions — Multiple Sclerosis; Stroke; Parkinson Disease; Brain Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- People with neurological disease according to inclusion criteria: People with neurological disease (Multiple Sclerosis, Parkinson Disease, Stroke and acquired brain injuries) will be recruited according to inclusion and exclusion criteria.
  Interventions: Device: Robotic Assisted Gait Training with G-EO system

INTERVENTIONS:
Device: Robotic Assisted Gait Training with G-EO system — Robotic-assisted gait training is a rehabilitation treatment that applies robotic technologies to improve mobility of patients with stroke or other neurological disorders. In this study, participants will use the G-EO system robotic device according to the daily clinical practice of the Don Gnocchi Foundation.

SUMMARY:
The aim of this work is to elaborate a statistical model to predict the effectiveness of robotic treatment in subjects with neurological diseases. The model will be used to understand which subjects are most responsive to this type of treatment

DETAILED DESCRIPTION:
In recent years, robotic devices have been used to assist balance and gait rehabilitation of people with neurological disorders. In particular, the G-EO system (Reha Technology AG, Switzerland) is a robotic end-effector device guiding the movement of the feet. It is currently unclear which variables are the predictors of treatment success. Indeed, the effectiveness of the GEO treatment may depends on the characteristics of the treatment itself (instrumental parameters defined by the physiotherapist using the device) and on the characteristics of the subject receiving the treatment. Therefore, it is necessary to measure these clinical and instrumental characteristics to understand which are predictors of treatment effects. Parameters obtained from this assessment can be used to elaborate statistical models. In our study the statistical model will be defined as follows: The change in the primary outcome measure after the robotic treatment will be considered as dependent variable of the model. All the "secondary" clinical outcome measures will be measured only at T0 and will be considered in the model as independent variables, along with the participants characteristics (age, gender, disease, disease duration, falls number, numbers of comorbidity, type of hospitalization) and the treatment characteristics (sessions number, frequency, duration, step length, cadence, gait speed, body weight support, distance traveled). The results of the model will suggest which subjects are most responsive to this type of treatment and which variables can be considered as predictors of the treatment success.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Multiple Sclerosis, Parkinson Disease, Stroke or acquired brain injury
* Minimum number of sessions: 10 sessions with the GEO system
* Minimum frequency of sessions: 2 per week
* Age ≥ 18 years
* Ability to walk for at least 10 meters, also with aid
* Indication of robotic treatment in the therapeutic plan
* Body size suitable for the robotic device
* ability to maintain verticality for 7 minutes;
* ability to maintain the sitting position without support for 30 seconds;

Exclusion Criteria:

* severe limitations of articular range of motion;
* medical problems compromising walking (e.g. fractures, pain, severe osteoporosis or severe spasticity);
* Presence of skin lesions in the areas of contact with the device;
* Presence of seizures that may be triggered by the use of the G-EO system.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People with Neurological Disease, in particular people with Multiple Sclerosis (MS), Parkinson Disease (PD) and Stroke
Sampling Method: Non-Probability Sample
Enrollment: 260 (Estimated)
Dates: Start 2022-05-13 (Actual); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Change in gait speed | baseline (T0), at the end of the treatment in accordance with the duration foreseen by the therapeutic plan of each subject up to a minimum of 2 weeks, (T1) and 2 months of follow up
  The 10 Meter Walk Test is a performance measure used to assess walking speed in meters per second over a short distance.
  The time to cover 6 meters is measured and the walking speed is calculated. higher speed indicates better performance.

SECONDARY OUTCOMES:
Trunk control | baseline (T0)
  The Trunk Control Test can be used to assess the motor impairment of the trunk in a patient, the total score range is 0 (minimum) to 100 (maximum, indicating better performance)
Mobility | baseline (T0)
  The Modified Rivermead Mobility Index (MRMI) is recommended to assess mobility in neurological patients. the total score range is 0 (minimum) to 40 (maximum, indicating better mobility)
Strength | baseline (T0)
  The 5 time sit to stand test asses functional lower extremity strength, transitional movements, balance, and fall risk in older adults and patient population. The time to stand up and sit down 5 times is measured. Lower time indicates better performance.
Walking Endurance | baseline (T0)
  The 6 Minute Walk Test is a sub-maximal exercise test used to assess aerobic capacity and endurance. The distance covered over a time of 6 minutes is used as the outcome by which to compare changes in performance capacity. the distance covered in 6 minutes is measured. Greater distance indicates better performance.
Walking ability | baseline (T0)
  The modified Dynamic Gait Index (mDGI) measures the capacity to adapt gait to complex tasks utilizing 8 tasks and 3 facets of performance. The total score range is 0 (minimum) to 64 (maximum, indicating better performance)
Activities of daily living | baseline (T0)
  The Modified Barthel Index (MBI) is a Measure of physical disability used widely to assess behaviour relating to activities of daily living for stroke patients or patients with other disabling conditions. The total score range is 0 (minimum) to 100 (maximum, indicating no assistance required to complete daily activities)
Cognitive function | baseline (T0)
  The Frontal Assessment Battery (FAB) is a brief tool that can be used at the bedside or in a clinic setting to assist in discriminating between dementias with a frontal dysexecutive phenotype and Dementia of Alzheimer"s Type. The total score range is 0 (minimum) to 18 (maximum, indicating better performance)
Balance confidence | baseline (T0)
  The Activities-specific Balance confidence (ABC) scale is a questionnaire developed to assess older individual's balance confidence in performing daily activities. ABC scale consists of a wide continuum of less and more challenging daily activities. The total score range is 0 (minimum) to 100 (maximum, indicating better balance confidence in daily activities)
Community integration | baseline (T0)
  The Community Integration Questionnaire (CIQ) is a tool used by researchers to gather information about how connected people are to their communities.
  The total score range is 0 (minimum) to 29 (maximum, indicating greater integration)
Gait symmetry (Instrumental index) | baseline T0
  Symmetry index of the gait cycle in the AnteroPosterior plan. Higher indexes indicate better performance.
Gait regularity (Instrumental index) | baseline T0
  Regularity index of the gait cycle in the AnteroPoserior plan. Higher indexes indicate better performance.

CONTACTS AND LOCATIONS:
Locations (1):
- Don Gnocchi Foundation, Milan, Italy